CLINICAL TRIAL: NCT05951010
Title: Comparison of Two Therapeutic Approaches of Cerebellar Transcranial Direct Current Stimulation in a Sardinian Family Affected by Spinocerebellar Ataxia 38: a Clinical and Computerized 3D Gait Analysis Study.
Brief Title: Cerebellar Transcranial Direct Current Stimulation in Spinocerebellar Ataxia 38
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Collaborators: Angela Sanna (Unknown); Micaela Porta (Unknown); Paolo Tacconi (Unknown); Chiara Pau (Unknown)
Responsible Party: Principal Investigator, Massimiliano Pau, Full Professor of Bioengineering, University of Cagliari
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: tDCS-ATX
Record Dates: First submitted 2023-07-04; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Spinocerebellar Ataxias
Keywords: gait; ataxic symptoms; dysarthric symptoms
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial direct current stimulation (tDCS) (Experimental): Participants underwent anodal stimulation delivered by a battery-driven stimulator (Neuroelectrics, Barcellona, Spain) through a pair of saline-soaked surface sponge electrodes (7 x 5 cm2) producing a constant current of 2 mA for 20 min.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Anodal stimulation was delivered by a battery-driven stimulator (Neuroelectrics, Barcellona, Spain) through a pair of saline-soaked surface sponge electrodes (7 x 5 cm2) producing a constant current of 2 mA for 20 min. The anode was placed 2 cm under the inion and the cathode was placed over the right deltoid muscle (CD-tDCS) or the spinal lumbar enlargement (2 cm under T11) as described by Benussi et al. (CS-tDCS). An electroconductive gel was applied to the electrodes to reduce contact impedance and the electrodes were held in place using elastic gauzes.

SUMMARY:
Spinocerebellar ataxia 38 (SCA 38) is a very rare autosomal dominant inherited disorder caused by a mutation in ELOV5 gene, specifically expressed in cerebellar Purkinje cells, encoding an enzyme involved in the synthesis of fatty acids. The present study aimed to assess the effect of cerebellar anodal transcranial direct current stimulation (tDCS) administered employing deltoid (CD-tDCS) and spinal (CS-tDCS) cathodal montage. Clinical evaluation was performed at baseline (T0), after 15 sessions of tDCS (T1) and after one month of follow-up (T2).

ELIGIBILITY:
Inclusion Criteria:

1. age ≤ 80 and > 18 years
2. diagnosis of SCA 38 with the presence of clinical symptoms.

Exclusion Criteria:

1. Inability to understand and sign the informed consent
2. Presence of other severe neurological disorders
3. presence of significant medical or psychiatric illnesses
4. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Modified International Cooperative Ataxia Rating Scale (MICARS) | Baseline, change after 3 weeks, change after 3 months
  Modified International Cooperative Ataxia Rating Scale (MICARS) was used to rate ataxic symptoms. Scores range from 0 (no impairment) to 100 (maximum impairment) Higher scores indicate worse impairments
Robertson dysarthria profile | Baseline, change after 3 weeks, change after 3 months
  A clinical-perceptual method exploring all components potentially involved in speech difficulties. Minimum score is 0 (higher impairment) maximum score is 284 (no impairments) Higher scores indicate better speech abilties

SECONDARY OUTCOMES:
Gait Speed | Baseline, change after 3 weeks, change after 3 months
  Instrumental assessment of gait speed (m/s) using motion capture system. Higher speed indicate improvements
Step width | Baseline, change after 3 weeks, change after 3 months
  Instrumental assessment of step width (m) using motion capture system. Smaller values of step width indicate gait improvements
Double support phase duration | Baseline, change after 3 weeks, change after 3 months
  Instrumental assessment of double support phase duration (s) using motion capture system. Smaller values of double support phase duration indicate a more stable gait

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorio di Biomeccanica ed Ergonomia industriale - Università degli Studi di Cagliari, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanna A, Pau M, Pilia G, Porta M, Casu G, Secci V, Cartella E, Demattia A, Firinu S, Pau C, Milia A, Cocco E, Tacconi P. Comparison of Two Therapeutic Approaches of Cerebellar Transcranial Direct Current Stimulation in a Sardinian Family Affected by Spinocerebellar Ataxia 38: a Clinical and Computerized 3D Gait Analysis Study. Cerebellum. 2024 Jun;23(3):973-980. doi: 10.1007/s12311-023-01590-w. Epub 2023 Aug 4. PMID 37540312